CLINICAL TRIAL: NCT04195516
Title: The Effect of Health Promotion Program Applied to University Students on Improving Healthy Nutrition and Physical Activity Behaviors
Brief Title: Improving Healthy Nutrition and Physical Activity Behaviors of University Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: aysedost
Record Dates: First submitted 2019-08-20; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-08

CONDITIONS: Obesity; Students
Keywords: health promotion; university students; obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Promotion Group (Experimental): Experimental group will be applied Health Promotion Model Basic Health Promotion Program. Health promotion program; The Web-based Health Promotion Program includes individual counseling and reminder practices.
  Interventions: Other: web based training,individual counseling, using reminders
- Control Group (No Intervention): The control group will be given educational brochures to develop healthy eating and physical activity behaviors.

INTERVENTIONS:
Other: web based training,individual counseling, using reminders — Health Promotion Model based Health Promotion Program will be applied to the experimental group. Health promotion program; The Web-based Health Promotion Program includes individual counseling and reminder practices.
  Within the context of the Web Based Health Promotion Program, 8 weeks of training to improve healthy eating and physical activity behaviors, individual counseling will be given.
  Colorful picture reminders will be sent to the experimental group through Whatsapp groups.
  At the end of the intervention, cognitive and physical measurements of the students will be done at 1st, 3rd and 6th months.
  Arms: Health Promotion Group

SUMMARY:
There are many descriptive studies in the literature on health behaviors of university youth.However, there are a limited number of model-based interventional studies explaining the development of positive health behaviors of students in the university period.In this context, this study "Applied to University Students The aim of this study will be to determine the Impact of Health Promotion Program on Developing Healthy Nutrition and Physical Activity Behaviors.This study was planned as a randomized controlled experimental study to determine the effect of the health promotion program applied to university students on the development of healthy eating and physical activity behaviors. The general population of the study will be composed of students enrolled in a formal education program at Istanbul Medipol University between January and September 2019.

The study population will consist of students with a body mass index between 25-35 kg / m², a mean nutritional behavior score of 2 or less, no regular physical activity, and no musculoskeletal, cardiopulmonary, metabolic or other systemic problems that prevent exercise.The sample size was calculated by power analysis. In the calculation, 0,80 power value, 0,05 error level, 0,60 'relationship is predicted, sampling 45 students to the experiment, 45 students to the control group was found to be appropriate. Experimental and control groups will be appointed by making probable selection from the study universe. In the study process, 10 substitutes were selected considering that there could be subjects who could leave the research. After all; 55 people in the experimental group and 55 people in the control group were selected by sampling. The sample consisted of 110 students.

DETAILED DESCRIPTION:
1. In order to identify the risky students in the study universe, a stand will be opened in the most crowded area and the most frequently used area of the campus.
2. As a result of the screening, body mass indexes are between 25-35 kg / m², nutritional behavior score is 2 or less, do not perform regular physical activity and do not have problems related to musculoskeletal system, cardiopulmonary system, metabolic system and other systems. Students will be admitted to the study universe.
3. Assignment will be made to the experimental and control groups by making probable selection from the study population.
4. Measurements of physical and cognitive variables of experimental and control groups will be made.
5. Health Promotion Modeled Health Promotion Program (Annex-1) will be applied to the experimental group. Health promotion program; The Web-based Health Promotion Program includes individual counseling and reminder practices. The content of the Web Based Health Promotion Program is given in Annex-2. The control group will be given educational brochures to develop healthy eating and physical activity behaviors.
6. Measurements of physical and cognitive variables of experimental and control groups at 1st, 3rd and 6th months will be made.
7. The data will be analyzed and evaluated statistically.
8. Report will be written.

ELIGIBILITY:
Inclusion Criteria:

Students with body mass indexes between 25-35 kg / m² Nutritional behavior of students with a mean score of 2 and below Students who do not do regular physical activity

Exclusion Criteria:

Students who have problems with musculoskeletal system, cardiopulmonary system, metabolic system and other systems that will prevent exercise will not be accepted.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
physical activity variables | start, 1st, 3rd, 6th month
  Post-intervention BMI and weight average of students participating in health promotion model based health promotion program will be lower than pre-program and non-program group.

SECONDARY OUTCOMES:
nutrition behaviors variables | start, 1st, 3rd, 6th month
  The average number of meals consumed by the students who participated in the health promotion model based health promotion program after the initiative will be higher than the pre-program and non-program group.
nutrition behaviors variables-2 | start, 1st, 3rd, 6th month
  The daily drinking water amount of students participating in the health promotion model based health promotion program will be higher than the pre-program and non-program group.
physical activity variables-2 | start, 1st, 3rd, 6th month
  The average number of weekly steps of students participating in the health promotion model based health promotion program will be higher than the pre-program and non-program group.
nutrition behaviors variables-3 | start, 1st, 3rd, 6th month
  The average carbohydrate consumption consumed by the students participating in the health promotion model based health promotion program will be lower than the pre-program and non-program group consumed.
physical activity variables-3 | start, 1st, 3rd, 6th month
  International Physical Activity Questionnaire (IPAQ) score of students participating in health promotion model based health promotion program will be higher than pre-program and non-program group.
physical activity variables-4 | start, 1st, 3rd, 6th month
  Healthy Lifestyle Behaviors Scale Nutrition subscale score of students participating in health promotion model based health promotion program will be higher than pre-program and non-program group.
cognitive variables | start, 1st, 3rd, 6th month
  Self-efficacy Scale for Regulation of Nutritional Habits of students participating in health promotion model-based health promotion program will be higher than pre-program and non-program group.
cognitive variables-2 | start, 1st, 3rd, 6th month
  Self-efficacy Scale for Regular Exercise Scale of students participating in health promotion model-based health promotion program will be higher than pre-program and non-program group.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Dost, Lecturer, Principal Investigator — Medipol University; Melek Nihal Esin, Professor, Study Director — Istanbul University
Locations (1):
- İstanbul Medipol Üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
publish in international journals write a chapter in this field
Supporting Information: Study Protocol
Time Frame: after June 2020
Access Criteria: all person

REFERENCES:
- [Background] Napolitano MA, Whiteley JA, Mavredes MN, Faro J, DiPietro L, Hayman LL, Neighbors CJ, Simmens S. Using social media to deliver weight loss programming to young adults: Design and rationale for the Healthy Body Healthy U (HBHU) trial. Contemp Clin Trials. 2017 Sep;60:1-13. doi: 10.1016/j.cct.2017.06.007. Epub 2017 Jun 10. PMID 28611007
- [Background] Patrick K, Marshall SJ, Davila EP, Kolodziejczyk JK, Fowler JH, Calfas KJ, Huang JS, Rock CL, Griswold WG, Gupta A, Merchant G, Norman GJ, Raab F, Donohue MC, Fogg BJ, Robinson TN. Design and implementation of a randomized controlled social and mobile weight loss trial for young adults (project SMART). Contemp Clin Trials. 2014 Jan;37(1):10-8. doi: 10.1016/j.cct.2013.11.001. Epub 2013 Nov 9. PMID 24215774

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04195516/Prot_SAP_000.pdf
  • Informed Consent Form (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT04195516/ICF_001.pdf